CLINICAL TRIAL: NCT01986647
Title: On the Move: Optimizing Participation in Group Exercise to Prevent Walking Difficulty in At-Risk Older Adults
Brief Title: On the Move: Optimizing Participation in Group Exercise
Acronym: OTM-PCORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jennifer S. Brach, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO13090264
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Physical Disability
Keywords: exercise; older adults; mobility disability
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- On the Move Exercise - exercise leader (Experimental): On the Move group exercise - 2 times per week for 12 weeks. Each session lasts approximately 1 hour. Timing and coordination exercises to improve walking. Led by exercise leader
  Interventions: Behavioral: On the Move exercise - exercise leader
- Standard program - exercise leader (Active Comparator): Standard impairment based seated group exercise program. 2 times per week for 12 weeks, approximately 1 hour class. Led by exercise leader
  Interventions: Behavioral: Standard program - exercise leader
- On the Move - staff activity personnel (Active Comparator): On the Move group exercise - 2 times per week for 12 weeks. Each session lasts approximately 1 hour. Timing and coordination exercises to improve walking. Led by activity personnel.
  Interventions: Behavioral: On the Move exercise - staff activity personnel
- Standard - staff activity personnel (Active Comparator): Standard impairment based seated group exercise program. 2 times per week for 12 weeks, approximately 1 hour class. Led by staff activity personnel
  Interventions: Behavioral: Standard program - staff activity personnel

INTERVENTIONS:
Behavioral: On the Move exercise - exercise leader — exercise physiologists
  Arms: On the Move Exercise - exercise leader
Behavioral: Standard program - exercise leader — This is an impairment-based exercise program focusing on flexibility, strength and endurance and is taught by research staff who are PTs, PTAs, or exercise physiologists
  Arms: Standard program - exercise leader
Behavioral: On the Move exercise - staff activity personnel — this is a group exercise program focusing on the timing and coordination of walking. The program is taught by a person from the facility that the research team trained.
  Arms: On the Move - staff activity personnel
Behavioral: Standard program - staff activity personnel — This is an impairment-based exercise program focusing on flexibility, strength and endurance and is taught by a member of the facility that the research staff trained.
  Arms: Standard - staff activity personnel

SUMMARY:
Community-dwelling older adults fear loss of independence and nursing home placement more than death. Walking difficulty often leads to loss of independence. Exercise is beneficial to physical and mental health and may prevent walking difficulty and promote independence. Recognizing the importance of exercise, senior housing facilities offer exercise programs to their residents. The exercise programs are often group-based, seated range of motion exercises that do not challenge the older adult; consequently participation rates and resident satisfaction are low.

If the goal is to improve walking to promote independence than the exercise program should specifically target walking. Therefore, we developed a challenging, group exercise program entitled "On the Move" which focuses on the fundamentals of walking. In this research study we will determine if the On the Move program is better than a standard program at improving walking and promoting independence and if the same benefits can be obtained if the On the Move program is delivered by staff of the senior living facilities instead of an exercise leader. To answer these questions, 400 community-dwelling older adults living in 32 different Independent Living Facilities and Senior High Rises or living in the community and attending senior community centers will be randomly assigned to either the 12 week On the Move group exercise program or the standard group exercise program delivered by either an exercise leader or staff activity personnel. Participants' walking and reported ability to carry out everyday activities (functional ability) will be assessed before and after the 12 week program. We will also assess participant safety and satisfaction with the exercise program and instructor.

The findings from this research study will provide evidence for the value of the On the Move group exercise program and will better inform patient choices regarding participation in exercise programs. If successful in improving walking and promoting independence and acceptable to the older adult, the On the Move program could be incorporated into exercise programming for older adults in community centers, health clubs, and senior residences across the country.

DETAILED DESCRIPTION:
This single-blinded cluster randomized trial compares the effectiveness and sustainability of On the Move and a standard group exercise program in 400 community-dwelling older adults. We will also examine the acceptability and risks associated with exercise participation. We will accomplish the objectives by pursuing the following specific aims:

1. Compare the effects of the On the Move group exercise program to a standard program on self-reported function and disability and walking ability. The On the Move program will produce greater gains in self-reported function and disability (Late Life Function and Disability Index/LLFDI) and walking ability (6-minute walk test/6MWT and gait speed) when delivered by an exercise leader.
2. When feasible to be delivered by staff activity personnel, explore the effectiveness of On the Move compared to a standard program; and sustainability compared to delivery by exercise leaders (when feasible). Explore barriers to identifying and training staff activity personnel. On the Move delivered by staff activity personnel (when feasible) will produce gains in above outcomes that are greater than the standard program; and comparable to when delivered by an exercise leader.
3. Compare the acceptability and the risks of the On the Move and standard exercise programs delivered by (a) exercise leaders and (b) staff activity personnel (when feasible). On the Move will result in greater satisfaction and higher attendance rates than the standard program. Attendance rates and satisfaction will be similar for exercise leader and staff activity personnel led programs when feasible to recruit staff personnel. Adverse event (falls, soft tissue injuries, muscle soreness, etc) rates during exercise will be similar between the two groups and the two facilitators when feasible to recruit staff personnel.
4. Explore potential baseline predictors of benefit and risks of participation in On the Move program to facilitate informed patient decision making. We will be able to identify combinations of baseline physical, psychosocial and demographic factors associated with each of the treatment response and adverse events outcomes.

This single-blinded cluster randomized trial targets community-dwelling older adults residing in Independent Living Facilities and Senior High Rises or living in the community and attending senior community centers. The trial compares type of exercise program (12 week standard group exercise program to the 12 week On the Move group exercise program) and the mode of delivery (exercise leader to staff activity personnel). Primary outcomes include function, disability and walking ability. We will also examine acceptability and risks associated with exercise participation.

Study population We will recruit participants from the Independent Living Facilities (ILFs), Senior Housing sites and from senior community centers.

Interventions:

Exercise program comparison. The On the Move exercise program will be compared to a standard group exercise program. Both exercise programs will be group-based and led by a person. Both programs will be delivered by trained exercise leaders or trained staff activity personnel (only when such a person is available). When a suitable staff activity person is not available, the program will be delivered by one of our exercise leaders. The frequency and duration of the programs are identical (50 minutes, 2 times a week for 12 weeks). The main difference between the standard and the On the Move group exercise programs is the program content which is described below.

The On the Move exercise program is based on principles of motor learning that enhance "skill" or smooth and automatic movement control. The program contains a warm-up (5 minutes), stepping patterns (15 minutes), walking patterns (15 minutes), strengthening exercises (10 minutes), and cool-down exercises (5 minutes). The warm-up and cool down contain gentle range of motion exercises and stretches for the lower extremities and trunk. The stepping and walking patterns are goal-oriented progressively more difficult patterns which promote the timing and coordination of stepping, integrated with the phases of the gait cycle. The strengthening exercises are conducted in sitting and standing and target the lower extremity muscles. The majority of the program will be conducted in standing (40 minutes) with only a small portion conducted in sitting (10 minutes).

The standard group exercise program is based on exercise programs that are currently being conducted at the facilities (i.e. standard of care). The operationally defined program contains a warm-up (5 minutes), upper and lower extremity strength and flexibility exercises (30 minutes), static balance exercises (10 minutes) and a cool-down (5 minutes). The majority of the program will be conducted in sitting (40 minutes) with only a small portion (10 minutes) conducted in standing.

Sustainability of the program: exercise leader and staff activity personnel comparison (Aim 2). The sustainability of the program will be evaluated by assessing the effectiveness of On the Move compared to a standard program when delivered by staff activity personnel and by comparing outcomes obtained by the On the Move program delivered by exercise leaders and staff activity personnel.

Outcomes:

Our main outcomes, function, disability, and walking ability are highly associated with independence and are extremely important to the older adult. Our primary measure of function and disability is the Late Life Function and Disability Instrument (LLFDI) and our main measures of walking ability are Six Minute Walk Test (6MWT) and gait speed. We will also examine confidence in walking (Gait Efficacy Scale), walking under challenging conditions (challenging gait tasks and figure of 8 walk), and gait variability as additional measures of walking ability. All measures will be collected at baseline and immediately following the 12 week intervention by research personnel who are blinded to the intervention group assignment. All testing will be conducted at the ILFs and Senior Housing sites.

Data analysis:

Aim 1:

First, we will perform a multivariate Hotelling t-test to simultaneously compare the baseline to follow-up change in the three primary outcomes between the arms to protect the type I error rate from multiplicity. If significant, subsequent analyses will be performed without further multiplicity adjustment. If not, subsequent comparisons will be performed with a conservative Bonferroni correction at the α=0.05/4=0.0125 level. This protected test approach has been recommended in the statistical literature and used in other exercise intervention trials with multiple outcomes.

Second, we will fit a series of linear mixed models using the SAS® MIXED procedure with baseline to follow-up change in each of the continuous outcomes (LLFDI function/disability, walking ability, other measures of mobility performance) as the dependent variable; intervention arm (standard/On the Move), as the fixed effect of primary interest; baseline value of outcome as an additional fixed effect covariate; and a facility random effect to account for greater similarity of participants from the same facility compared to different facilities and resulting non-independence of observations within facility (ie. clustering). We will construct appropriate means contrasts to estimate difference in gains in the two interventions when delivered by exercise leaders (Aim 1) whose statistical significance of the estimates will serve as formal tests of hypotheses. We will consider adding other baseline measures found to be significantly different between the arms or deemed important as additional fixed effect covariates in the model to assess robustness of the findings. We note that waiting of participants randomized to staff activity personnel classes constitute a group of control participants, if smaller, without any intervention. Therefore, we will perform another sensitivity analysis employing a similar analytic strategy but with three intervention arms (On the Move/Standard/Wait List Control).

Aim 3(a):

We will fit a series of generalized estimating equations (GEE) models(68) using the SAS® GENMOD procedure with each of the dichotomous adverse events, adherence (21+ sessions or ≥90%) and satisfaction outcomes as the dependent variable; a binomial distribution for the outcome and a logit canonical link function; intervention arm, as the effect of primary interest; baseline value of outcome and any other measures found to be different between arms or deemed important as additional fixed effects covariates; and an exchangeable working correlation structure to account for clustering due to facility. We will appropriately construct contrasts to test hypotheses of differential proportions with adverse events based on intervention when delivered by exercise leaders.

Aims 2, 3(b) and 4 Exploratory Analyses

Aim 2:

We propose an analytic strategy with an exploratory philosophy for Aim 2 sustainability aim, because of the uncertainty surrounding our ability to recruit and train a staff activity person to lead a class safely and per protocol.

We will fit a series of linear mixed models using the SAS® MIXED procedure with baseline to follow-up change in each of the continuous outcomes (LLFDI function/disability, walking ability, other measures of mobility performance) as the dependent variable; intervention arm (standard/On the Move), delivery mode (by exercise leader/staff activity personnel) and their interaction as fixed effects of interest; baseline value of outcome and any other measures found to be different between arms or deemed important as additional fixed effects covariates; and a facility random effect to account for greater similarity of participants from the same facility compared to different facilities and resulting non-independence of observations within facility (ie. clustering). We will construct appropriate means contrasts to estimate difference in gains in the two interventions when delivered by staff exercise personnel (Aim 2 effectiveness hypothesis); and difference in gains attributable to On the Move intervention when delivered by exercise leaders and staff activity personnel (Aim 2 sustainability hypothesis). Statistical significance of the estimates will serve as formal tests hypotheses. We note that participants randomized to staff activity personnel had to wait 12 weeks since their baseline assessment and randomization to start the intervention, during which they may have changed; and that they underwent a second baseline assessment immediately prior to starting the exercise intervention. Therefore, we will repeat the above analysis using their second baseline assessment instead of the first one to assess the sensitivity of results.

Aim 3(b):

We will fit a series of generalized estimating equations (GEE) models using the SAS® GENMOD procedure with each of the dichotomous adverse events, adherence (21+ sessions or ≥90%) and satisfaction outcomes as the dependent variable; a binomial distribution for the outcome and a logit canonical link function; intervention arm, delivery model and their interaction as effects of interest; baseline value of outcome and any other measures found to be different between arms or deemed important as additional fixed effects covariates; and an exchangeable working correlation structure to account for clustering due to facility. We will appropriately construct contrasts to test hypotheses of differential proportions with adverse events based on intervention when delivered by staff activity personnel and delivery mode.

Aim 4:

We will perform the exploratory analyses to identify combinations of baseline predictors of treatment response and risks of participating in On the Move program.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* resident of University of Pittsburgh Medical Center Independent Living Facility or senior housing site
* Ambulate independently for household distance (may use a straight cane)

Exclusion Criteria:

* non English speaking
* impaired cognition defined as unable to follow 2 step commands
* plans to leave area in next 4 months
* progressive neuromuscular disorder
* any acute illness or medical condition that is not stable
* inappropriate response on 6 minute walk test

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 424 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Brach, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Brach JS, Perera S, Gilmore S, VanSwearingen JM, Brodine D, Wert D, Nadkarni NK, Ricci E. Stakeholder involvement in the design of a patient-centered comparative effectiveness trial of the "On the Move" group exercise program in community-dwelling older adults. Contemp Clin Trials. 2016 Sep;50:135-42. doi: 10.1016/j.cct.2016.08.003. Epub 2016 Aug 10. PMID 27521806
- [Derived] Coyle PC, Perera S, Albert SM, Freburger JK, VanSwearingen JM, Brach JS. Potential long-term impact of "On The Move" group-exercise program on falls and healthcare utilization in older adults: an exploratory analysis of a randomized controlled trial. BMC Geriatr. 2020 Mar 16;20(1):105. doi: 10.1186/s12877-020-1506-3. PMID 32178633
- [Derived] Brach JS, Perera S, Gilmore S, VanSwearingen JM, Brodine D, Nadkarni NK, Ricci E. Effectiveness of a Timing and Coordination Group Exercise Program to Improve Mobility in Community-Dwelling Older Adults: A Randomized Clinical Trial. JAMA Intern Med. 2017 Oct 1;177(10):1437-1444. doi: 10.1001/jamainternmed.2017.3609. PMID 28806436

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 2014 through January 2016. Potential participants were recruited from independent living facilities, senior apartment buildings, and senior community centers.
Groups:
- On the Move Exercise Group - Exercise Leader: On the Move group exercise - 2 times per week for 12 weeks. Each session lasts approximately 1 hour. Timing and coordination exercises to improve walking. Taught by exercise leader.
  On the Move group exercise
- Standard Group Exercise Program - Exercise Leader: Standard impairment based seated group exercise program. 2 times per week for 12 weeks, approximately 1 hour class. Taught by exercise leader
  Standard group exercise
- On the Move Exercise Program - Staff Activity Personnel: On the Move group exercise - taught by staff activity personnel
- Standard Exercise Program - Staff Activity Personnel: Standard exercise program taught by a member of the facility who does not necessarily have formal exercise training. this person will be trained by the research staff to lead the class.
  Standard group exercise
Period: Overall Study
Arm/Group | On the Move Exercise Group - Exercise Leader | Standard Group Exercise Program - Exercise Leader | On the Move Exercise Program - Staff Activity Personnel | Standard Exercise Program - Staff Activity Personnel
Started | 152 | 146 | 49 | 77
Completed | 142 | 139 | 37 | 66
Not Completed | 10 | 7 | 12 | 11
Not completed — Lost to Follow-up | 4 | 1 | 4 | 4
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 3
Not completed — Health | 5 | 3 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- On the Move Exercise Group - Exercise LEader: On the Move group exercise - 2 times per week for 12 weeks. Each session lasts approximately 1 hour. Timing and coordination exercises to improve walking.
  Exercise class will be led by a person who is trained in exercise such as exercise physiologist, physical therapist, physical therapist assistant On the Move group exercise
- Standard Group Exercise Program - Exercise Leader: Standard impairment based seated group exercise program. 2 times per week for 12 weeks, approximately 1 hour class.
  Exercise class will be led by a person who is trained in exercise such as exercise physiologist, physical therapist, physical therapist assistant Standard group exercise
- On the Move Group - STaff Activity Personnel: On the Move group exercise - 2 times per week for 12 weeks. Each session lasts approximately 1 hour. Timing and coordination exercises to improve walking.
  Exercise class will be led by a member of the facility who does not necessarily have formal exercise training. this person will be trained by the research staff to lead the class.
  On the Move group exercise
- Standard Program - Staff Activity Personnel: Standard impairment based seated group exercise program. 2 times per week for 12 weeks, approximately 1 hour class.
  Exercise class will be led by a member of the facility who does not necessarily have formal exercise training. this person will be trained by the research staff to lead the class.
  Standard group exercise
- Total: Total of all reporting groups
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel | Total
Number analyzed (Participants) | 152 | 146 | 49 | 77 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.6 (8.2) | 80.5 (8.1) | 83.7 (6.2) | 81.7 (7.0) | 80.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 120 | 40 | 58 | 349
  Male | 21 | 26 | 9 | 19 | 75
Region of Enrollment [Number; unit: participants]
  United States | 152 | 146 | 49 | 77 | 424
Intervention Setting [Count of Participants; unit: Participants]
  Community center | 36 | 29 | 13 | 14 | 92
  Independent living facility | 42 | 61 | 29 | 44 | 176
  Apartment building | 74 | 56 | 7 | 19 | 156
Married [Count of Participants; unit: Participants] | 29 | 30 | 22 | 18 | 99
College education [Count of Participants; unit: Participants] | 67 | 73 | 28 | 47 | 215
Comorbidities [Mean (Standard Deviation); unit: units on a scale] — Measured using the Duke Comorbidity Index. The scale asks if a doctor ever told you that you have XXXXXX? The items are consolidated into systems impacted. Scores range from 0-8 with 8 indicating a greater disease burden.
  units on a scale | 2.9 (1.4) | 2.7 (1.5) | 2.8 (1.3) | 3.0 (1.3) | 2.8 (1.4)
Fear of falling [Count of Participants; unit: Participants] | 53 | 57 | 17 | 21 | 148
fall in previous year [Count of Participants; unit: Participants] | 45 | 41 | 16 | 26 | 128
Excellent/Very good mobility [Count of Participants; unit: Participants] | 90 | 90 | 30 | 37 | 247
Excellent/very good health [Count of Participants; unit: Participants] | 80 | 75 | 32 | 38 | 225
Excellent/very good balance [Count of Participants; unit: Participants] | 47 | 51 | 14 | 19 | 131
Height [Mean (Standard Deviation); unit: meters] | 1.61 (0.10) | 1.61 (0.13) | 1.6 (0.2) | 1.6 (0.1) | 1.6 (0.12)
Weight [Mean (Standard Deviation); unit: kg] | 75.3 (21.1) | 71.9 (15.7) | 74.1 (32.0) | 74.3 (18.0) | 73.8 (20.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.03 (7.59) | 28.62 (15.76) | 31.4 (24.3) | 27.6 (6.1) | 28.9 (13.4)
Six minute walk distance [Mean (Standard Deviation); unit: meters] | 273.3 (88.0) | 277.3 (95.5) | 276.2 (88.7) | 282.8 (82.6) | 276.8 (89.6)
LLFDI function [Mean (Standard Deviation); unit: units on a scale] — Late Life Function and Disability Instrument, Function scale Scores range 0-100 with a greater score indicating better function.
  units on a scale | 58.9 (8.5) | 60.0 (10.5) | 59.6 (8.6) | 59.8 (9.5) | 59.5 (9.4)
LLFDI disability [Mean (Standard Deviation); unit: units on a scale] — Late Life Function and Disability Instrument - Disability component. Scores range from 0-100 with a greater score indicating less disability.
  units on a scale | 53.3 (6.5) | 51.6 (5.8) | 54.0 (6.6) | 52.6 (6.7) | 52.7 (6.4)
Gait speed [Mean (Standard Deviation); unit: m/s] | 0.90 (0.20) | 0.92 (0.21) | 0.91 (0.18) | 0.91 (0.20) | 0.92 (0.21)

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-reported Overall Function From Baseline to 12 Weeks
Description: Late Life Function and Disability Index (LLFDI) overall function. Scores range from 0-100 with higher score representing better function.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | On the Move Exercise Group - Exercise Leader | Standard Group Exercise Program - Exercise Leader | On the Move Exercise Program - Staff Activity Personnel | Standard Exercise Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
units on a scale | 0.4 (5.7) | -0.6 (5.8) | -1.37 (4.68) | -0.32 (6.03)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise Leader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.2691, Mixed Models Analysis; linear mixed model due to clustering by facility and multiple imputation for missing data

2. Primary Outcome: Change in Self-reported Disability From Baseline to 12 Weeks
Description: Late Life Function and Disability Instrument (LLFDI) disability frequency component. Scores range from 0-100 with higher scores representing better (less) disability.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
units on a scale | 0.4 (4.1) | 0.7 (5.0) | -1.45 (6.34) | 1.26 (5.66)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.6087, Mixed Models Analysis; linear mixed model due to clustering by facility and multiple imputation for missing data

3. Primary Outcome: Change in Gait Speed From Baseline to 12 Weeks
Description: Gait speed in m/s
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: m/s
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
m/s | 0.05 (0.13) | -0.01 (0.11) | -0.01 (0.13) | 0.02 (0.16)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; linear mixed model due to clustering by facility and multiple imputation for missing data

4. Primary Outcome: Change in Six Minute Walk Distance From Baseline to 12 Weeks
Description: distance walked in 6 minutes
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: meters
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
meters | 20.6 (57.1) | 4.1 (55.6) | 9.3 (72.4) | -3.24 (56.48)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.0344, Mixed Models Analysis; linear mixed model due to clustering by facility and multiple imputation for missing data

5. Secondary Outcome: Number of Participants Who Reported They Benefited a Good Bit or Somewhat From the Class
Description: Participant satisfaction will be measured by satisfaction surveys and personal interviews. Benefited from class a good bit or somewhat
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
Participants | 104 | 105 | 21 | 41
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.6879, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.49 to 1.60]

6. Secondary Outcome: Number of Participants Who Reported That the Class Was at Least Somewhat Challenging
Description: Measured by question on the satisfaction questionnaire. Question asked participants to rate how challenging the class was.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
Participants | 92 | 94 | 23 | 33
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.5719, Regression, Logistic; Risk Difference (RD) = 0.88, 95% CI 2-sided [0.56 to 1.37]

7. Secondary Outcome: Number of Participants Reporting That They Received a Just Right Amount of Individualized Instruction
Description: Question from satisfaction questionnaire - that asked participants their opinion on the amount of individualized instruction they received.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
Participants | 128 | 124 | 25 | 53
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.489, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.44 to 5.53]

8. Secondary Outcome: Number of Participants Who Reported That They Felt Safe or Very Safe During the Exercise.
Description: Question from the satisfaction questionnaire.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
Participants | 131 | 127 | 27 | 58
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.2981, Regression, Logistic; Odds Ratio (OR) = 3.12, 95% CI 2-sided [0.37 to 26.6]

9. Secondary Outcome: Number of Participants Who Reported They Were Satisfied or Very Satisfied With the Program.
Description: Question from the satisfaction questionnaire.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
Participants | 128 | 126 | 26 | 57
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.9279, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.30 to 3.74]

10. Secondary Outcome: Number of Participants Who Reported They Would Definitely or Probably Continue With the Program
Description: Question from the satisfaction questionnaire.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
Participants | 113 | 108 | 26 | 56
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.5835, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.67 to 2.06]

11. Secondary Outcome: Change in Figure 8 Walk Test From Baseline to 12 Weeks
Description: Time it takes to walk a figure 8 around 2 cones 5 feet apart. Greater time in seconds represents poorer performance
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | On the Move Exercise Group - Exercise Leader | Standard Group Exercise Program - Exercise Leader | On the Move Exercise Program - Staff Activity Personnel | Standard Exercise Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
seconds | -0.67 (2.02) | 0.11 (3.15) | -0.1 (2.1) | 0.3 (3.9)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise Leader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.18, Mixed Models Analysis; Mean Difference (Final Values) = -0.64, Standard Error of Mean 0.46

12. Secondary Outcome: Change in Modified Gait Efficacy Scale From Baseline to 12 Weeks
Description: Confidence in walking was measured by the modified gait efficacy scale (mGES). Scores range from 0-100 with higher scores indicating greater confidence.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
units on a scale | -0.61 (10.7) | -1.51 (12.1) | -5.3 (11.6) | -4.1 (11.5)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.73, Mixed Models Analysis; Mean Difference (Final Values) = 0.51, Standard Error of Mean 1.42

13. Secondary Outcome: Change in Short Physical Performance Battery From Baseline to 12weeks
Description: Short physical Performance Battery is a performance test that includes gait speed, 5 time sit to stand and standing balance. Scores range from 0-12 with greater scores indicating better performance.
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
units on a scale | 0.16 (1.81) | 0.17 (1.53) | -0.1 (2.4) | -0.1 (1.7)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.71, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, Standard Error of Mean 0.28

14. Secondary Outcome: Change in Stance Time Variability From Baseline to 12weeks
Description: variability of individual stance times during walking as measured from a electronic walkway. Measured as the standard deviation of all stance times. greater values represent greater variability which is related to poorer outcomes.
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
seconds | 0.002 (0.03) | 0.00 (0.03) | 0.006 (0.02) | -0.001 (0.022)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.77, Mixed Models Analysis; Mean Difference (Final Values) = 0.001, Standard Error of Mean 0.004

15. Secondary Outcome: Change in Narrow Walk Time From Baseline to 12 Weeks
Description: Time to walk narrow pathway. Greater values (times) indicate poorer performance.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
seconds | -0.25 (2.04) | -0.04 (2.39) | -0.3 (1.5) | 0.1 (2.6)
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.80, Mixed Models Analysis; Mean Difference (Final Values) = -0.11, Standard Error of Mean 0.44

16. Other Pre Specified Outcome: Attendance Rates
Description: The number of participants attending 20 or more exercise classes
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | On the Move Exercise Group - Exercise LEader | Standard Group Exercise Program - Exercise Leader | On the Move Group - STaff Activity Personnel | Standard Program - Staff Activity Personnel
Number analyzed (Participants) | 152 | 146 | 49 | 77
Participants | 76 | 95 | 12 | 40
Statistical Analysis 1: Comparison: On the Move Exercise Group - Exercise LEader vs Standard Group Exercise Program - Exercise Leader; Test type: Superiority or Other; p = 0.0324, Regression, Logistic; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.29 to 0.95]

ADVERSE EVENTS:
Arm/Group | On the Move Exercise - Exercise Leader | Standard Program - Exercise Leader | On the Move - Staff Activity Personnel | Standard - Staff Activity Personnel
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/146 | 0/49 | 1/77
Other Adverse Events (participants affected / at risk) | 4/152 | 0/146 | 2/49 | 0/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On the Move Exercise - Exercise Leader (N=152) | Standard Program - Exercise Leader (N=146) | On the Move - Staff Activity Personnel (N=49) | Standard - Staff Activity Personnel (N=77)
chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — participant experienced chest pain during the exercise class. participant had a history of cardiovascular disease.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On the Move Exercise - Exercise Leader (N=152) | Standard Program - Exercise Leader (N=146) | On the Move - Staff Activity Personnel (N=49) | Standard - Staff Activity Personnel (N=77)
fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — fall during the exercise class
pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fatigue (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No